CLINICAL TRIAL: NCT06352710
Title: Determining Postoperative Recovery and the Impact of Adverse Events in Neurosurgery Based on Self-reported, App-based Longitudinal Assessment - a Collaborative Observational Research Project
Status: Recruiting | Type: Observational
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Alexis P. R. Terrapon, MD, Cantonal Hospital of St. Gallen
Other Study IDs: 2022-01510
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Disc Disease; Instabilities Lumbar; Brain Tumor; Aneurysm
Keywords: Outcome; PROMs; App; Neurosurgery; Adverse event; Complication; Quality of life; TDN
MeSH Terms: conditions — Brain Neoplasms; Aneurysm; Alzheimer Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Lumbar decompression, including single- or multiple-level procedures
  Interventions: Other: OP-Tracker App
- Lumbar transpedicular instrumentation and fusion, including extension to thorax/pelvis
  Interventions: Other: OP-Tracker App
- Supratentorial craniotomy for tumor, vascular or other pathology
  Interventions: Other: OP-Tracker App
- Infratentorial craniotomy for tumor, vascular or other pathology
  Interventions: Other: OP-Tracker App

INTERVENTIONS:
Other: OP-Tracker App — There will be no study-specific therapeutic intervention. The OP-Tracker App will be downloaded and installed on the patient's smartphone. Preoperative assessment: baseline factors such as age, gender, medical conditions, type of disease and of surgery, EQ-5D-5L. Before and after surgery surgery, SWI (Quality of life) will be assessed daily using "pop-ups"; the patient will input the value (0-10) using a slide-bar. After completion of the surgery, the app will automatically modify the number of SWI assessments over time according to the occurrence of AEs. At any point in time, the patient will be able to register an AE in the smartphone app. The patient can select the AE via a drop-down menu in the app, and can additionally input free text in case of an AE of type "other". Using a further drop-down menu, the patient will classify the AE according to the CDG and TDN grade. QoL assessments (EQ-5D-5L questionnaire) will pop up before, and at 3 and 12 months after surgery.

SUMMARY:
Analyzing the impact of surgery and adverse events (AEs) on patients' well-being is of paramount importance as it provides essential information for benefit-risk assessment. Current methods in outcome research are static, resource-intensive and subject to missing-data issues. Moreover, AEs are inconsistently reported using various grading systems that usually do not account for patients' subjective well-being. These are severe drawbacks for outcome research as it hinders monitoring, comparison, and improvement of treatment quality.

The increasing use of smartphones offers unprecedented opportunities for data collection. We developed a free smartphone application to assess fluctuations of patients' well-being as a result of surgical treatment and possible AEs. The application is installed on each patient's smartphone and collects standardized data at defined timepoints before and after surgery (well-being, AE description and severity).

By acquiring longitudinal patient-reported outcome before and after neurosurgical interventions, we aim to determine the regular postoperative course for specific surgical procedures, as well as any deviation thereof, depending on the occurrence and severity of AEs. We will evaluate the validity of existing AE classifications and, if necessary, propose a new patient-centered scheme. We hope that this will result in an increase in standardized reporting of patient outcome, and ultimately allow for evidence-based patient information and decision-making.

DETAILED DESCRIPTION:
Understanding and analyzing the impact of surgery and adverse events (AEs) on the subjective well-being of patients is of paramount importance as it provides objective information that may be useful in a risk-benefit discussion. Current methods in outcome research are static, resource-intensive and subject to missing-data issues. This results in a poor understanding of the normal postoperative course which in turn prevents consistent reporting of AEs as they are usually defined as a deviation thereof. As an additional challenge and because there is no consensus and/or recommendation on this subject, AEs are graded using various classifications that neglect the impact of AEs on the subjective well-being of patients. For example, the most used AE grading system is the therapy-based Clavien-Dindo-Grading system (CDG, doi:10.1097/01.sla.0000133083.54934.ae), which fails to detect the severity of AE that are not treated by means of pharmacotherapy and/or surgery. This is an important limitation as new neurologic deficits are frequent AEs that may imply dramatic consequences on quality of life but are considered as low grade in therapy-based grading systems such as the CDG. Other classifications were developed specifically for neurosurgery but they suffer the same limitations. Recently, our group proposed the Therapy-Disability-Neurology Grade (TDN, doi:10.1093/neuros/nyab121) to address this problem. The TDN grade takes into account the therapy used to counteract AEs (as does the CDG), the associated neurologic deficits, and the resulting disability, but currently lacks widespread use and validation. These are severe drawbacks for outcome research as it hinders monitoring, comparison, and improvement of quality of the treatment delivered.

The increasing use of smartphones across all age groups offers unprecedented opportunities for data collection. We have created a smartphone application (app) to assess patient well-being in a standardized and longitudinal fashion. The app named "Op-tracker app". It collects longitudinal, self-reported data (subjective well-being rated from 0 to 10) at fixed time points before and after surgery. Additional information such as type of disease, type of surgery (currently four categories), AE description and severity (according to the CDG and TDN grade) is also recorded, along with a standardized quality of life (QoL) questionnaire (EQ-5D-5L). A simplified version recently described in a feasibility study showed good acceptance and no major technical issues (doi:10.1007/s00701-021-04967-0). With this innovative technique of data acquisition, we will gather a higher density of data using less resources than traditional methods.

In a prospective observational pilot study without intervention using the "op-tracker app" to acquire longitudinal patient reported outcome measures (the subjective well-being index, SWI) before and after surgery, we aim to determine the regular postoperative course for certain surgical procedures as well as the deviation thereof depending on the severity of specific AEs. We will evaluate the validity of existing AE severity grading systems and if necessary, propose a classification more consistent with the subjective well-being of patients. This will greatly benefit patient information by providing essential insight about standard and complicated postoperative course. Beyond the benefit this new data will add to the scientific literature, we hope that the app will improve daily patient care by enabling early detection of and reaction to AEs in case of "pathological decrease" in self-reported well-being and QoL. Should this be confirmed, the app could be widely used and its scope could be extended to the whole neurosurgical spectrum or even to further surgical subspecialties. We anticipate that this will result in an increase in standardized reporting of patient outcome and ultimately in a more evidence-based patient information and decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* The patient must be able to consent
* The patient is willing to provide data upon one year after surgery
* The patient possesses and is capable of using a smartphone (Android or iOS operative systems)
* The patient has the necessary language and cognitive skills to use the smartphone app
* The patient is scheduled for one of the defined operations (see above for both spinal and cranial) and in a stable, non-life-threatening situation (admitted to the regular ward or intermediate care unit (IMC))
* Baseline preoperative SWI and QoL assessment is possible (minimum requirement is one assessment, the latest the day before surgery)

Exclusion Criteria:

* Pregnancy
* Foreseeable difficulties using the smartphone or smartphone app
* The presence of a condition that hinders the baseline preoperative assessment
* Health conditions that render inclusion unsafe (e.g., untreated ruptured intracranial aneurysm or congestive heart failure; in general, all patients admitted to the intensive care unit (ICU))

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing either one of the defined non-urgent surgical interventions on the neurocranium or the spine interested in participating in this study will be considered. Patients admitted urgently will only be considered if the surgery is not performed on the day of hospital admission, to allow for the baseline evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2025-06-12 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Subjective Well-Being (SWI) | Until 2 years after study begin
  The variable of primary interest is a patient reported outcome measure (PROM), the SWI, expressing the subjective well-being of patients from 0 to 10. To describe the regular postoperative course (SWI variation) after each type of surgical procedure (and according to baseline variables such as age, gender, underlying pathology, comorbidities), as well as the deviation thereof in patients who experience an AE, we will use (Generalized) Linear Mixed-effects Models (GLMMs).

SECONDARY OUTCOMES:
EQ-5D-5L | Until 2 years after study begin
  The difference in standardized QoL questionnaire (EQ-5D-5L) [14] before as compared to 3 and 12 months after an operation (as well as sub-analysis for each type of surgery and with vs without an AE).
Rate of adverse events | Until 2 years after study begin
  The difference in the rate of AEs in the first year after surgery between different types of surgery.
Severity of adverse events | Until 2 years after study begin
  The difference in the distribution of the severity (using the CDG and TDN grade) of AEs in the first year after surgery between different types of surgery.
Correlation between TDN/CDG and SWI/QoL | Until 2 years after study begin
  The correlation between the severity of AEs in the first year after surgery (using the CDG system and the TDN grade) and postoperative SWI and QoL (EQ-5D-5L).
Correlation between baseline factors and TDN grade | Until 2 years after study begin
  The relationship between patient-specific variables (e.g., age, sex, etc.) and the rate as well as severity of AEs in the first year after surgery.
Difference between rate of adverse events and TDN distribution between different surgery groups | Until 2 years after study begin
  The difference in the rate and severity of AEs in the first year after surgery for different groups of patients (for example according to underlying pathology, other medical conditions, or a combination of such factors).

CONTACTS AND LOCATIONS:
Locations (1):
- Kantonsspital St.Gallen, Sankt Gallen, Switzerland